CLINICAL TRIAL: NCT04367597
Title: A Roll-over Study of CM-2019 Trial (A Randomized, Sham Controlled, Double-blind, Multi-center Study of Neuromuscular Electrical Stimulation (NMES) as an Adjunctive Therapy for Knee Pain Relief and Improving Functional Outcomes in Knee Osteoarthritis (OA) Patients)
Brief Title: Evaluation of NMES Therapy for Pain Relief Associated With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CyMedica Orthopedics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM-2019R
Record Dates: First submitted 2020-04-23; First posted 2020-04-29 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized, sham-controlled, double-blind, multi-center
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active NMES (Experimental)
  Interventions: Device: Home-based Neuromuscular Electrical Stimulation (NMES) therapy
- Modified NMES sham (Sham Comparator)
  Interventions: Device: Home-based Neuromuscular Electrical Stimulation (NMES) therapy

INTERVENTIONS:
Device: Home-based Neuromuscular Electrical Stimulation (NMES) therapy — A home-based NMES treatment applied by the subjects daily

SUMMARY:
A roll-over study of the current CM-2019 trial to assess the same preplanned outcomes of CM-2019 at 14 weeks.

DETAILED DESCRIPTION:
This roll-over study is designed as a 14-week treatment continuation from CM-2019 (parent study), a randomized, sham controlled, double-blind, multi-center study trial to evaluate the efficacy of CyMedica Orthopedics e-vive™ system, a multifunctional electrotherapy device providing neuromuscular electrical stimulation (NMES) as an adjunctive therapy for pain relief and accelerating functional recovery in patients with knee osteoarthritis. This follow-up trial will include subjects who have been randomized into the CM-2019 trial. Subjects will be enrolled into the appropriate treatment group based upon the treatment received in the parent study. It is hypothesized that the continued use of CyMedica e-vive NMES may provide additional pain relief and improved knee function for an additional 14 weeks compared to sham.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide a signed informed consent for CM-2019R. The subject will be provided with a copy of the signed Informed Consent upon signature.
2. Currently enrolled in the parent trial CM-2019 or have successfully completed the parent trial within 21 days of enrollment in the roll-over trial.
3. Willing and able to continue parent trial study treatment.
4. Pregnancy test, if it has been >14 days since completion of the parent trial.
5. Subject must continue to be willing to refrain from receiving knee intra-articular injections of steroids, knee intra-articular injections of hyaluronic acid, opioids, and analgesics (except for acetaminophen up to 3000 mg/day or an equivalent) for the duration of the study.
6. Subject must continue to be willing to take acetaminophen (up to 3000 mg/day) or an equivalent as pain medication for the duration of the study.
7. Subject must continue to be willing to stop taking any pain medications 24 hours prior any scheduled study visit.
8. Subject must continue to be willing to stop receiving knee physical therapy of the target knee for the duration of the study.
9. Subject must continue be willing to stop wearing any knee unloader brace of the target knee for the duration of the study.
10. Subjects must be willing and able to comply with all study procedures for the duration of the clinical study

Exclusion Criteria:

1. Subjects with a new diagnosis of inflammatory arthritis (knee rheumatoid arthritis, active gout, knee joint infection, Lyme disease, SLE, etc.) since parent trial enrollment.
2. Subjects with a new diagnosis of severe neuropathy condition and under medication for treatment of the condition since parent trial enrollment.
3. Subjects with a new diagnosis of fibromyalgia since parent trial enrollment.
4. Subjects who have had an injury or an acute traumatic injury to the target knee since parent trial enrollment.
5. Subject must NOT have had arthroscopy of the target knee since parent trial enrollment.
6. Subjects who have had treatment of the target knee with intra-articular injections of steroids since parent trial enrollment. Subjects who have had intra-articular injections of hyaluronic acid since parent trial enrollment.
7. Subjects who have a scheduled surgery on the target knee within the study period. (Subjects that are contemplating the surgery can be included.)
8. Subjects who have used electrotherapy or acupuncture for OA of the target knee since parent trial enrollment year.
9. Subjects who have had implanted electrical devices since parent trial enrollment (cardiac pacemakers, deep brain stimulators, implantable cardiac defibrillators).
10. Subjects with a current new malignancy or who have received treatment for malignancy since parent trial enrollment, with the exception of resected basal cell carcinoma and squamous cell carcinoma of the skin.
11. Subjects with a new skin breakdown or infection in the area where the study device will be placed (quadriceps of the target knee).
12. Subjects with any newly reported chronic conditions (e.g., diabetes, hypertension, congestive heart failure, etc.) or that have not been well-controlled during the parent trial.
13. Subjects who have any new litigation for worker's compensation.
14. Subjects with any new condition, in the opinion of the Investigator that might interfere with the evaluation of the study objectives.
15. Subjects who are pregnant.
16. Subject who enrolled in any new clinical study from the last day of treatment in the parent trial that required the use of an investigational device, drug or biologic.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Knee pain | 14 weeks post intervention
  Assessment of knee pain relief associated with knee osteoarthritis using VAS instrument scale
Knee pain and function | 14 weeks post intervention
  Assessment of knee pain relief and function improvements associated with knee osteoarthritis using WOMAC survey
Knee pain and function | 14 weeks post intervention
  Assessment of knee pain relief and function improvements associated with knee osteoarthritis using KOOS Jr. survey

SECONDARY OUTCOMES:
Knee function | 14 weeks post intervention
  Knee functional improvements including quadriceps strength tes
Knee function | 14 weeks post intervention
  Knee functional improvements including Timed Up and Go test
Knee function | 14 weeks post intervention
  Knee functional improvements including 3 Min walk test
Knee function | 14 weeks post intervention
  Knee functional improvements including Repeated chair rise test

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Noble Clinical Research, Tucson, Arizona
  - Tucson Orthopedic Institute, Tucson, Arizona
  - Synergy Group US LLC, Houston, Texas
  - Synergy Group US LLC, Katy, Texas
  - Synergy Group US LLC, Missouri City, Texas

IPD SHARING:
Plan to Share IPD: No